CLINICAL TRIAL: NCT05772403
Title: Contrast-enhanced Ultrasound (CEUS) Improves Characterization of Atypical Liver Nodules in Patients With Chronic Liver Disease
Brief Title: Contrast Enhanced Ultrasound (CEUS) in Atypical Liver Nodules in Patients With Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4288
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CEUS — CEUS for atypical liver nodules

SUMMARY:
The present study aims to investigate the role of CEUS in evaluating liver lesions with atypical characteristics on contrast-enhanced CT or MRI. All patients enrolled in the study underwent contrast-enhanced ultrasound. Based on CEUS characteristics, atypical nodules will be categorized according to CEUS LI-RADS classification.

DETAILED DESCRIPTION:
This retrospective study investigates the role of CEUS in evaluating liver lesions with atypical characteristics on contrast-enhanced CT or MRI. All patients enrolled in the study underwent contrast-enhanced ultrasound. All CEUS exams were performed, recorded, and analyzed by two experienced operators (>10 years of experience with abdominal US and CEUS). Based on CEUS characteristics, atypical nodules will be categorized according to CEUS LI-RADS (LR) classification. If the analyzed nodule shows a typical hallmark on CEUS (LR-5), that is arterial phase hyperenhancement with late-onset (>60 s) washout of mild intensity, it is definitively considered HCC and have been treated appropriately. Categories LR-3 and LR-4 comprise nodules with different combinations of arterial and venous phase enhancement features, expected to correspond to an intermediate or high probability of lesions to be HCC. Patients with LR-3 or LR-4 nodules underwent follow-up; in some cases they underwent biopsy.

LR-M is used to classify high-probability malignant lesions but nonspecific for HCC; these nodules underwent biopsy for further characterization.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of liver cirrhosis or chronic liver disease with increased risk of HCC
* diagnosis of atypical nodules on contrast-enhanced CT or MRI

Exclusion Criteria:

* less than 18 years of age
* pregnancy
* typical nodules on contrast-enhanced CT or MRI
* non-visualized nodule on B-mode US
* CEUS not performed or performed more than three months after CT or MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for liver cirrhosis or chronic liver disease with increased risk of HCC (HBV-related hepatopathy or fibrosis F3) and diagnosed with liver atypical nodules on contrast-enhanced CT or MRI.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
The role of CEUS in evaluating atypic liver lesions on contrast-enhanced CT or MRI. | Between January 2018 and January 2023
  The primary endpoint is to assess the contrastographic behaviour of nodules suspected of HCC and defined as atypical by contrast-enhanced CT and MRI, using CEUS. Prevalence of CEUS LI-RADS categories among atypical nodules will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico A Gemelli Irccs, Roma, RM, Italy